CLINICAL TRIAL: NCT04403581
Title: Cross-sectional Descriptive Study: Egyptian Doctors Stresses, Knowledge and Attitude During COVID-19 Pandemic
Brief Title: Egyptian Doctors Stresses, Knowledge and Attitude During COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Riham H Raafat, Lecturer of Chest diseases, Ain Shams University
Other Study IDs: Egyptian doctors in COVID-19
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Covid-19
Keywords: stresses; covid-19; doctors
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — Questionnaire for assessing stresses, knowledge and attitudes of doctors in COVID-19 pandemic

SUMMARY:
Doctors are at high risk of corona virus infection (COVID-19) during pandemic. The investigators are aiming to explore the emotions, perceived stressors, knowledge and coping strategies of doctors who are working during COVID-19 pandemic in different specialties and in different hospitals by a self assessment questionnaire that was designed and modified from two previously published articles (mentioned in the references), including 7 sections with 88 questions.

DETAILED DESCRIPTION:
Background

Corona virus disease 2019 (COVID-19), an infectious respiratory disease caused by a newly discovered corona virus in December 2019, has been recognized as a serious threat to global health. Since the WHO declared COVID-19 a pandemic in early March 2020, the WHO and the Center for Disease Control and Prevention (CDC) have been considered the most reliable sources of information for the COVID-19 global pandemic. The CDC listed moderate to severe asthma, especially if not well controlled, as high-risk for severe illness from COVID-19.

A large number of cases occurred among health care workers (HCW), which were contracted within the health care facilities. Some of the HCWs even died from the COVID-19 disease. Moreover, it was reported that unrecognized, asymptomatic patients transferred to their family or close contacts. All these factors were alarming and potentially distressing for the hospital staff who worked during the pandemic.

The severe acute respiratory syndrome (SARS) epidemic in 2003 also involved disease transmission to HCWs. Even though the fatality rates for SARS were lower than for COVID-19 infection, nonetheless, they were a cause of significant stress, emotional turmoil, and concern for all the SARS healthcare providers.

The emotions, perceived stressors, complete knowledge assessment and coping strategies of HCWs especially doctors during COVID-19 have not been explored. These issues were the intended focus of the study.

ELIGIBILITY:
Inclusion Criteria:

* doctors from different specialties

Exclusion Criteria:

* doctors who stopped working in the pandemic

Ages: 23 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Working doctors in different specialties
Sampling Method: Non-Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Cross-sectional descriptive study: Egyptian Doctors Stresses, Knowledge and Attitude during COVID-19 Pandemic | 2 months
  Highlighting the emotional aspects, perceived stressors, level of knowledge and coping strategies of doctors who are working during COVID-19 pandemic in different hospitals by using questionnaires that the investigators gave the name "COVID-19 Doctor Stress Questionnaire" that included 7 sections with 88 questions:
  1. Demographic data related questions
  2. Doctors feelings related questions
  3. Factors that help in stressing doctors
  4. Factors help in reducing stresses
  5. Questions detecting knowledge
  6. Attitude towards stresses
  7. Motives to complete work Each is answered by the participant and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Riham H Raafat, MD, Principal Investigator — Ainshams university

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: World Health Organization. Pneumonia of unknown cause - China: disease outbreak news. Geneva:, January 5, 2020 — https://www.who.int/csr/don/05-january-2020-pneumonia-of-unkown-cause-china/en/
- See also: Oboho IK, Tomczyk SM, Al-Asmari AM, Banjar AA, Al-Mugti H, Aloraini MS, et al 2014 MERS-CoV outbreak in Jeddah--a link to health care facilities. N Engl J Med 2015; — https://pubmed.ncbi.nlm.nih.gov/25714162/
- See also: Lee SH, Juang YY, Su YJ, Lee HL, Lin YH, Chao CC. Facing SARS: psychological impacts on SARS team nurses and psychiatric services in a Taiwan general hospital. Gen Hosp Psychiatry 2005;27:352-358. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4851451/
- See also: Ahmed I. Albarraka,, Rafiuddin Mohammed, Ali Al Elayan, Feras Al Fawaz, Musab Al Masry, Mohammed Al Shammari, Saud Bin Miaygil: MERS: Comparing the knowledge, attitude and practices of different health care workers. — https://doi.org/10.1016/j.jiph.2019.06.029